CLINICAL TRIAL: NCT06976216
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Evaluate the Efficacy and Safety of KarXT + KarX-EC for the Treatment of Cognitive Impairment Associated With Mild to Moderate Alzheimer's Disease (MINDSET 1)
Brief Title: A Study to Evaluate the Efficacy and Safety of KarXT + KarX-EC for Cognitive Impairment in Alzheimer's Disease
Acronym: MINDSET 1
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CN012-0051; 2025-520746-30 (EudraCT Number); U1111-1317-4462 (Other: UTN)
Record Dates: First submitted 2025-05-09; First posted 2025-05-16 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Alzheimer's Disease
Keywords: Dementia; Cognitive Impairment; Kar-XT; KarX-EC; Mild Alzheimer's Disease; Moderate Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease; Dementia; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- KarXT + KarX-EC (Active Comparator)
  Interventions: Drug: KarXT; Drug: KarX-EC
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: KarXT — Specified dose on specified days
  Other Names: BMS-986510
  Arms: KarXT + KarX-EC
Drug: KarX-EC — Specified dose on specified days
  Other Names: BMS-986519
  Arms: KarXT + KarX-EC
Other: Placebo — Specified dose on specified days
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of KarXT + KarX-EC for cognitive impairment in Alzheimer's Disease

ELIGIBILITY:
Inclusion Criteria

* Participants must have a confirmed diagnosis of Alzheimer's disease (AD), specifically at the mild (stage 4) or moderate (stage 5) dementia stages, as defined by the National Institute on Aging and Alzheimer's Association (NIA-AA) core clinical criteria. The diagnosis of AD pathology must be confirmed through the 2024 revised NIA-AA Workgroup criteria using a stepwise diagnostic approach.
* Participants must have an Mini-Mental State Examination (MMSE) score ranging from 12 through 22, inclusive, at the time of screening.
* Participants must have a designated caregiver who maintains adequate contact (around 10 hours per week or more) and is willing to attend all study visits. The caregiver must also be responsible for reporting on the participant's condition, overseeing medication compliance, and consenting to their involvement in both their own and the participant's study-related activities.
* Participants on acetyl choline esterase inhibitors (AChEIs) and/or memantine, must have been on a stable dosage for at least 12 weeks prior to screening, and agree to maintain this stable dose for the study duration.

Exclusion Criteria

* Participants must not present with any significant or severe medical conditions that could compromise their safety, the ability to comply with or complete the study, or the integrity of the study results. This includes any grade of hepatic impairment, urinary retention, active biliary disease, moderate-severe renal impairment (eGFR of <50 mL/min), and unstable hypertension or tachycardia.
* Participants must not have any primary psychiatric diagnoses such as major depression, schizoaffective disorder, or bipolar disorder, and those with severe psychiatric symptoms that could complicate the interpretation of treatment effects, impair cognitive assessment, or impact study completion.
* Participants must not have a history of schizophrenia or other chronic psychosis, as well as those who have previously been exposed to KarXT or are currently undergoing treatment with disease-modifying anti-amyloid therapies for AD within the past 6 months prior to screening.
* Participants must not have significant pathological findings on brain magnetic resonance imaging (MRI) at screening that reflect significant pathology other than AD or could affect safety or interfere with study procedures.
* Other protocol-defined Inclusion/Exclusion criteria apply.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 586 (Estimated)
Dates: Start 2025-07-14 (Actual); Primary Completion 2028-09-11 (Estimated); Study Completion 2029-02-23 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Alzheimer's Disease Assessment Scale-Cognitive Subscale 11 (ADAS-Cog11) | At week 24
Clinician's Interview-Based Impression Plus Caregiver Input (CIBIC+) | At week 24

SECONDARY OUTCOMES:
Change from baseline in Alzheimer's Disease Cooperative Study-Activities of Daily Living scale (ADCS-ADL) | At week 24
Change from baseline in neuro psychiatric inventory (NPI) total score | At week 24
Number of participants with adverse events (AEs) | At week 24
Number of participants with serious adverse events (SAEs) | At week 24
Number of participants with adverse event of special interest (AESIs) | At week 24
Number of participants with AEs leading to study intervention discontinuation | At week 24
Number of participants with AEs leading to study discontinuation | At week 24
Number of participants with AEs leading to death | At week 24
Number of participants with clinically significant changes in vital signs | At week 24
Number of participants with clinically significant changes in electrocardiogram (ECG) tests | At week 24
Number of participants with clinically significant changes in Columbia-Suicide Severity Rating Scale (C-SSRS) tests | At week 24
Number of participants with clinically significant changes in weight | At week 24
Number of participants with clinically significant changes in safety laboratory tests | At week 24

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (111):
- United States (28):
  - Healthy Brain Clinic, Long Beach, California
  - Anderson Clinical Research, Redlands, California
  - Mountain Neurological Research Center, Basalt, Colorado
  - Local Institution - 0024, Washington D.C., District of Columbia
  - JEM Research Institute, Atlantis, Florida
  - VIN-Julie Schwartzbard, Aventura, Florida
  - Merritt Island Medical Research, LLC, Merritt Island, Florida
  - Renstar Medical Research, Ocala, Florida
  - Alzheimer's Research and Treatment Center, Stuart, Florida
  - Charter Research - Lady Lake, The Villages, Florida
  - Local Institution - 0016, Columbus, Georgia
  - Center for Advanced Research & Education, Gainesville, Georgia
  - Re:Cognition Health - Chicago, Chicago, Illinois
  - Ascension Alexian Brothers, Elk Grove Village, Illinois
  - Boston Center for Memory, Newton, Massachusetts
  - HealthPartners Neuroscience Center, Saint Paul, Minnesota
  - Advanced Memory Research Institute of New Jersey, Toms River, New Jersey
  - Local Institution - 0101, New York, New York
  - Local Institution - 0259, New York, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - AMC Research, LLC, Matthews, North Carolina
  - Ohio State University, Columbus, Ohio
  - Neurology Diagnostics, Inc., Dayton, Ohio
  - Summit Headlands, Portland, Oregon
  - Local Institution - 0004, Abington, Pennsylvania
  - Rhode Island Mood & Memory Research Institute, East Providence, Rhode Island
  - Neurology Clinic, P.C., Cordova, Tennessee
  - Gadolin Research, Beaumont, Texas
- Argentina (6):
  - Local Institution - 0088, Banfield, Buenos Aires
  - Local Institution - 0001, Buenos Aires, Buenos Aires F.D.
  - Local Institution - 0271, Buenos Aires
  - Local Institution - 0232, Córdoba
  - Sanatorio Morra S.A., Córdoba
  - Instituto Kremer, Córdoba
- Australia (5):
  - Local Institution - 0279, Kogarah, New South Wales
  - KARA Institute for Neurological Diseases, Macquarie Park, New South Wales
  - NeuroCentrix, Carlton, Victoria
  - Neurodegenerative Disorders Research, Perth, Western Australia
  - Local Institution - 0244, Darlinghurst
- Brazil (4):
  - Local Institution - 0168, Brasília, Federal District
  - Local Institution - 0180, Curitiba, Paraná
  - Local Institution - 0266, Aracaju, Sergipe
  - Hospital das Clinicas FMUSP, São Paulo
- Canada (8):
  - OCT Research ULC, Kelowna, British Columbia
  - Richmond Clinical Trials, Richmond, British Columbia
  - Centricity Research Halifax Multispecialty, Halifax, Nova Scotia
  - Ottawa Memory Clinic, Ottawa, Ontario
  - Toronto Memory Program, Toronto, Ontario
  - MoCA Research and Innovation Inc., Greenfield Park, Quebec
  - Diex Recherche Victoriaville, Victoriaville, Quebec
  - ALPHA Recherche Clinique, Québec
- Chile (5):
  - Local Institution - 0230, Antofagasta, AN
  - Local Institution - 0272, Providencia, Santiago Metropolitan
  - Local Institution - 0094, Santiago, Santiago Metropolitan
  - Local Institution - 0089, Santiago, Santiago Metropolitan
  - Local Institution - 0241, Santiago, Santiago Metropolitan
- Croatia (5):
  - Local Institution - 0215, Zagreb, City of Zagreb
  - Local Institution - 0284, Zagreb, City of Zagreb
  - Local Institution - 0216, Osijek
  - Local Institution - 0267, Rijeka
  - Local Institution - 0240, Zagreb
- Czechia (7):
  - Neuro Health Centrum, Brno, Brno-město
  - Local Institution - 0225, Olomouc, Olomoucký kraj
  - A-Shine, Pilsen, Plzeň-město
  - Neurologická Ambulance - Forbeli, Prague, Praha 6
  - Neuropsychiatrie, Prague, Praha 6
  - Local Institution - 0222, Prague, Praha 8
  - Vestra Clinics, Rychnov nad Kněžnou
- Germany (6):
  - TUM Klinikum, München, Bavaria
  - Local Institution - 0219, Münster, North Rhine-Westphalia
  - Local Institution - 0276, Mainz, Rhineland-Palatinate
  - Local Institution - 0218, Berlin
  - Local Institution - 0277, Bremen
  - Local Institution - 0275, Hamburg
- Greece (5):
  - Local Institution - 0281, Alexandroupoli, Anatolikí Makedonía Kai Thráki
  - Local Institution - 0256, Athens, Attikí
  - Aiginiteio University Hospital, Athens, Attikí
  - Local Institution - 0251, Thessaloniki, Thessaloníki
  - Local Institution - 0257, Larissa, Thessalía
- India (5):
  - Local Institution - 0288, Bengaluru, Karnataka
  - Local Institution - 0282, Hyderabad, Telangana
  - Local Institution - 0285, Hyderabad, Telangana
  - Local Institution - 0287, Varanasi, Uttar Pradesh
  - Local Institution - 0286, Kolkata, West Bengal
- Italy (4):
  - Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico, Milan, Lombardy
  - Ospedale San Raffaele, Milan, Lombardy
  - Local Institution - 0248, Monza, Lombardy
  - Azienda Ospedaliera Spedali Civili di Brescia, Brescia
- Poland (4):
  - Local Institution - 0262, Poznan, Greater Poland Voivodeship
  - Local Institution - 0261, Torun, Kuyavian-Pomeranian Voivodeship
  - Local Institution - 0280, Bialystok, Podlaskie Voivodeship
  - Centrum Badan Klinicznych PI-House sp. z o.o., Gdansk, Pomeranian Voivodeship
- Local Institution - 0181, San Juan, Puerto Rico
- Romania (5):
  - Local Institution - 0278, Bucharest, București
  - Local Institution - 0269, Bucharest, București
  - Local Institution - 0273, Bucharest, București
  - Prof. Dr. Alexandru Obregia Psychiatry Hospital, Bucharest, București
  - Local Institution - 0268, Iași
- South Korea (7):
  - Chonnam National University Hospital, Gwangju, Kwangju-Kwangyǒkshi
  - Seoul National University Bundang Hospital, Seongnam, Kyǒnggi-do
  - Seoul National University Hospital, Seoul, Seoul-teukbyeolsi [Seoul]
  - Hanyang University Seoul Hospital, Seoul, Seoul-teukbyeolsi [Seoul]
  - Konkuk University Medical Center, Seoul, Seoul-teukbyeolsi [Seoul]
  - Samsung Medical Center, Seoul, Seoul-teukbyeolsi [Seoul]
  - Ewha Womans University Seoul Hospital, Seoul, Seoul-teukbyeolsi [Seoul]
- Spain (6):
  - Hospital Victoria Eugenia, Seville, Andalusia
  - Hospital Universitari General de Catalunya, Sant Cugat del Vallès, Barcelona [Barcelona]
  - Hospital Clínic de Barcelona, Barcelona, Catalunya [Cataluña]
  - Hospital Universitari de Santa Maria, Lleida, Lleida [Lérida]
  - Clinica Universidad de Navarra, Pamplona, Navarre
  - Hospital Clinico San Carlos, Madrid

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT06976216.html